CLINICAL TRIAL: NCT01429142
Title: AIMS Study: Cost-effectiveness of a Nurse-based Intervention to Support HIV-treatment Adherence
Brief Title: AIMS Study: Improving HIV Treatment Adherence
Acronym: AIMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other); Maastricht University (Other)
Responsible Party: Principal Investigator, Marijn de Bruin, Professor, University of Aberdeen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AIMS_171002208
Record Dates: First submitted 2011-08-25; First posted 2011-09-05 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: HIV
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AIMS intervention (Experimental): see http://bmchealthservres.biomedcentral.com/articles/10.1186/1472-6963-13-274
  Interventions: Behavioral: AIMS intervention
- Treatment as usual (Active Comparator): see http://www.tandfonline.com/doi/abs/10.1080/08870446.2014.1001392
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Treatment as usual — In this multi-center trial, the content of usual adherence care is not known prior to the study, but it is part of our data collection to examine the content and variability between clinics and professionals afterwards.
  Arms: Treatment as usual
Behavioral: AIMS intervention — The AIMS-intervention is counseling intervention, using MEMS-data printed in simple plots. The following intervention steps will be followed:
  -Discussion of practical, tailored information about adherence -Identification of desired adherence level and motivations -Print of patients' MEMS-report and comparison with desired level -ID causes of non-adherence and how to deal with problems -Designing a tailored action plan. -Follow-up: evaluation of accomplishments, remaining problems and solutions, until desired level of adherence has been accomplished. -Formulation of goals for behavioral maintenance.
  Among patients starting treatment, the same elements will be delivered but MEMS-feedback can only be incorporated in the second session (after medication has been used). Moreover, a readiness element is added at treatment initiation, where patients discuss the necessity and concerns of initiating medication and are offered the possibility to practice intake for 2 weeks with placebo.
  Arms: AIMS intervention

SUMMARY:
The objectives of the main study are to evaluate the effectiveness and the cost-effectiveness of a counseling intervention to support medication intake among patients treated for HIV. The aim is that through the availability of medication intake reports collected through electronic monitoring, more adherence problems can be identified and medical decision-making improves.

A substudy focuses on the broader range of nursing care in HIV-treatment, examining the content of care delivered to support physical, mental, sexual and social well-being; whether the delivery of the AIMS intervention affects the quality of care on domains other than adherence; and whether the content of care on these various domains can be linked to patient well-being and satisfaction.

DETAILED DESCRIPTION:
**MAIN STUDY**

BACKGROUND: Adherence to HIV-medication is an important predictor of treatment success, yet between 25-40% of the patients does not always take the medication as prescribed. A nurse-delivered counseling intervention (AIMS: Adherence Improving self-Management Strategy) to optimize patient adherence has shown promising results in a pilot study and a randomized controlled trial among Caucasian, treatment-experienced patients. AIMS is a patient-centered counseling intervention to support self-regulation of medication intake, using feedback reports of electronically monitored adherence. AIMS has been evaluated positively by patients and nurses, and has been developed to be implemented in usual patient care against minimal time and monetary investments.

OBJECTIVE: To examine the cost-effectiveness of the AIMS intervention compared to "care-as-usual" in Dutch HIV-clinics among a representative sample of patients (all ethnicities, starting or already on treatment).

SETTING AND PARTICIPANTS: The study will be conducted in seven HIV-clinics in the Netherlands and select 230 patients (details regarding sample size calculation: see below) eligible for intervention based on the following criteria: 1- All treatment experienced patients who started combination AntiRetroviral Therapy (cART) ≥1996, are >9 months on treatment, are continuing treatment, and had at least one detectable viral load (blips included) during the last 3 years (count starts after 9 months cART). 2- All treatment-naïve patients initiating treatment.

After initial inclusion, treatment experienced patients with suboptimal adherence measured during a 2-month electronic monitoring baseline period will be eligible for randomization to the intervention or the control group. Treatment-initiating patients will be randomized directly after consenting.

DESIGN: A prospective multicenter trial with randomization of patients within nurses. Eligible treatment experienced patients with suboptimal adherence after 2 months baseline adherence monitoring will be randomized to receive either usual care plus the AIMS-intervention, or care as usual. Next, randomized experienced patients will visit the clinic every 4-5 months, with a minimum of 3 visits during at least a 15-month period (including the baseline period a total of 17 study months). Treatment-naïve patients will be randomized directly after consenting. As part of the AIMS-intervention, intervention participants are encouraged to start with a 2-week readiness trajectory before initiating cART. After initiating cART, control and intervention participants return for a visit after 2-4 weeks, 3-4 months, 6-7 months, 9-10 months, and 12-15 months.

PRIMARY MEASURES: Viral load, health care usage, quality of life, and adherence data will be obtained. MEMS-data will only be collected among half of the control group (randomly assigned to MEMS y/n).

OUTCOMES: 1- Primary cost-effectiveness outcome: a) costs per point increase in the proportion of patients with an undetectable viral load, b) costs per Quality Adjusted Life Year (QALY) gained. Secondary: Costs per one point increase in adherence as measured with the MEMS-caps.

2- Primary effectiveness outcome: The number of detectable viral loads at study months 6-7, 10-11, and 14-15 for experienced patients, and months 6-7, 9-10, and 12-15 for patients starting treatment. Secondary: Adherence according to MEMS-caps.

**PROJECT OBJECTIVES SUB STUDY** BACKGROUND: HIV-nurses' tasks go beyond discussing and supporting adherence, and include promoting patients' sexual, mental, physical and social well-being. Hence, it will be important to establish whether delivering the AIMS-intervention impacts the quality/scope of usual clinic care on these other important domains. In addition, measuring the content of usual care during the trial provides the opportunity to explore whether this is related to patients' well-being (sexual, mental, physical, social) and satisfaction with care.

OBJECTIVES: 1- To monitor the content of usual care on the different HIV-nursing domains and examine whether usual care content predicts patients' well-being and satisfaction with HIV-care at follow-up. 2- Explore whether delivering the AIMS-intervention has (dis)advantageous effects on the content and impact of usual care on domains other than adherence (sexual, mental, physical, social).

PARTICIPANTS: HIV-nurses and patients in the study clinics.

DESIGN AND MEASURES: HIV-nurses' usual care with regard to adherence, as well as mental, sexual, social and physical health will be assessed through questionnaires at randomization and at the end of the study. In addition, HIV-nurses will complete a brief online checklist after each study visit indicating the main topics discussed during that meeting. At randomization and after the study, patients will complete a brief questionnaire about their mental, social, physical and sexual health, and satisfaction with their care on these domains.

PRIMARY OUTCOMES: 1- The relation between the content of care with patient satisfaction and well-being. 2- Potential effects of AIMS on the content of care and patient well-being and treatment satisfaction.

SAMPLE SIZE CALCULATION:

During the initial grant application, a sample size was computed based on the assumption that only non-adherent, treatment experienced patients would be approached. However, following the input from participating clinics, the final inclusion and exclusion criteria were formulated as explained below. An updated sample size computation was done after inclusion had been initiated, which was submitted to (date: 27th February, 2013) and accepted by (date: 15th April, 2013) the funder (ZonMw, the Netherlands Organisation for Health Research and Development) using actual trial data in order to enhance accuracy of the estimates (the expected treatment effect is the same in both computations, the other estimates were adjusted to match then new criteria and available data).

Initial sample size calculation:

The sample size for the primary outcome measure was computed on the basis of a dichotomous dependent variable (detectable versus undetectable viral load), The data was planned to be analyzed using a multi-level model (patients nested within nurses) that would account for differential intervention effects between nurses. A total sample of 432 patients (18 nurses) was required to detect significant intervention effects at post-intervention with an alpha = .05 (two-sided) and 80% power, based on the following assumptions: depending on the nurse, (a) 60% to 80% of the patients have an undetectable viral load during usual care (i.e. ≥ 6 months after start of cART), (b) this increases in the intervention condition compared to the control condition by 5 to 20 percentage points, and (c) a nurse recruits on average 25 patients for the trial. (d) We expected a maximum dropout of 20%. We therefore intended to include 450 patients.

Updated sample size calculation:

The updated sample size computation is the following: A sample of 230 patients (22 nurses) is required to obtain 80% power to detect a significant intervention effect on viral load for at least one of three time points (for treatment-experienced patients: T1, T2, and T3; for treatment-initiating patients: T3, T4, and T5) with alpha=.05 (two-sided) and using a Bonferroni correction. Viral load at baseline is used as a covariate. A multilevel model is used with random intercepts and random treatment effects at the nurse level. The sample size calculation is based on the following assumptions: depending on the nurse, (a) 60% to 80% of treatment-initiating patients have an undetectable viral load during usual care (i.e. ≥ 6 months after start of ART), (b) 15% to 20% of treatment experienced-patients and all treatment-initiating patients have a detectable viral load at baseline, (c) this increases in the intervention condition compared to the control condition by 5 to 20 percentage points, (d) a nurse recruits on average 11 patients for the trial, and (e) an expected maximum dropout of 10%.

ELIGIBILITY:
Inclusion Criteria treatment-naive patients initiating cART:

- All patients are eligible

Inclusion criteria treatment experienced patients:

* Started cART after 1996, and
* Have been on cART for at least 9 months, and
* Had at least one detectable viral load (including blips) during the last 3 years (counting of these 3 years starts after the first 9 months on cART), and
* Had suboptimal adherence (<95% BID, <100% QD) during 2 months baseline measurement.

Exclusion criteria for treatment-naive and experienced patients:

* Age <18 years
* Psychiatric disorders or other comorbidities precluding compliance with study procedures
* Pregnancy
* Plans to interrupt treatment in the next 14 months
* Life expectancy less than one year as determined by physician
* Not able to communicate in English or Dutch
* HIV resistant to three or more of the currently available antiretroviral drug classes
* About to initiate intensive hepatitis C treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2011-09; Primary Completion 2014-06 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Cost-effectiveness: Costs per point increase in viral load | Month 0-14
  The costs and savings over the whole intervention period (post randomization until end of study) will be weighed against any gains observed in viral load (continuous or dichotomous: see primary effectiveness outcomes).
Effectiveness: Viral load | Month 4-14
  The combined viral load at 3 pre-determined time points after the initial intervention phase will serve as the primary outcome measure. Depending on the distribution, data will be kept continuous (log transformed) or recoded to detectable versus undetectable. Planned measurements naive patients at 6-7 months, 9-10 months, and 12-14 months post-randomization. For treatment experienced patients: 4-5 months, 8-10 months, and 12-15 months after randomization.

SECONDARY OUTCOMES:
Cost-effectiveness: Costs per point increase in adherence | Month 0-14
  The costs and benefits of intervention versus control care during the study will be weighed against any improvements in adherence following the initial intervention stage. For that purpose, adherence data during follow-up (i.e. the last 4 months of the study) will be used.
Cost-effectiveness: Costs per quality adjusted life year gained | month 0-14
  The costs and benefits of the intervention versus control care will be weighed against any differences observed in quality of life measured at 3 time points following the initial intervention period (time points are the same as for the primary effectiveness outcome)
Effectiveness: Adherence | Month 0-4, Month 5-8, Month 9-12
  Repeated measures analyses on adherence. Time windows will show some variation due to treatment stage of patient and clinic variation, but stratification and cluster randomization should prevent unequal distribution over groups.

CONTACTS AND LOCATIONS:
Overall Officials: Jan M Prins, PhD, Principal Investigator — Academic Medical Center - University of Amsterdam (AMC-UVA); Marijn de Bruin, PhD, Principal Investigator — University of Aberdeen
Locations (7):
- Netherlands (7):
  - Erasmus Medical Center, Rotterdam, South Holland
  - Sint Lucas Andreas Ziekenhuis, Amsterdam
  - Slotervaartziekenhuis, Amsterdam
  - Academic Medical Center, Amsterdam
  - Leiden Universitair MEdisch Centrum, Leidern
  - Haga Ziekenhuis, location Leyweg, The Hague
  - Isala Klinieken, Zwolle

IPD SHARING:
Plan to Share IPD: Yes
Upon request

REFERENCES:
- [Derived] Wijnen BFM, Oberje EJM, Evers SMAA, Prins JM, Nobel HE, van Nieuwkoop C, Veenstra J, Pijnappel FJ, Kroon FP, van Zonneveld L, van Hulzen AGW, van Broekhuizen M, de Bruin M. Cost-effectiveness and Cost-utility of the Adherence Improving Self-management Strategy in Human Immunodeficiency Virus Care: A Trial-based Economic Evaluation. Clin Infect Dis. 2019 Feb 1;68(4):658-667. doi: 10.1093/cid/ciy553. PMID 30239629
- [Derived] de Bruin M, Oberje EJM, Viechtbauer W, Nobel HE, Hiligsmann M, van Nieuwkoop C, Veenstra J, Pijnappel FJ, Kroon FP, van Zonneveld L, Groeneveld PHP, van Broekhuizen M, Evers SMAA, Prins JM. Effectiveness and cost-effectiveness of a nurse-delivered intervention to improve adherence to treatment for HIV: a pragmatic, multicentre, open-label, randomised clinical trial. Lancet Infect Dis. 2017 Jun;17(6):595-604. doi: 10.1016/S1473-3099(16)30534-5. Epub 2017 Mar 3. PMID 28262598
- [Derived] Oberje E, de Bruin M, Evers S, Viechtbauer W, Nobel HE, Schaalma H, McCambridge J, Gras L, Tousset E, Prins J. Cost-effectiveness of a nurse-based intervention (AIMS) to improve adherence among HIV-infected patients: design of a multi-centre randomised controlled trial. BMC Health Serv Res. 2013 Jul 17;13:274. doi: 10.1186/1472-6963-13-274. PMID 24059292